CLINICAL TRIAL: NCT01121679
Title: French Observatory on Hospitalizations in Cardiology of Patients of 80 Years and Over
Acronym: OCTOCARDIO
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Moubarak Ghassan, Assistant Professor, French Cardiology Society
Other Study IDs: 09472
Record Dates: First submitted 2010-04-16; First posted 2010-05-12 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Disease
Keywords: Older patients; Aged, 80 and Over; Cardiology
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients aged 80 years and older: Patients aged 80 years and older and hospitalized in a cardiology department

SUMMARY:
Because of increased life expectancy and improved therapeutic methods in cardiology, the proportion of very old patients with cardiovascular disease increases. However, clinical practice "in real life" are still insufficiently known in this population. The recommendations still lack of studies specifically devoted to elderly or very elderly, an extrapolation of data based on evidence obtained in younger populations.

This is a multicenter observational study during a day. On this day, all participating centers fill a questionnaire for each patient 80 years or older hospitalized in their service.

DETAILED DESCRIPTION:
Information about the center will be collected: non-university or university center, presence of coronary angiography room, number of beds, number of patients 80 years or older hospitalized in the day of the investigation.

The questionnaire is designed to:

* Know the history of cardiovascular and noncardiovascular patient and degree of dependence
* Know the reason for hospitalization
* Evaluate the diagnostic and therapeutic already implemented or planned for this patient

The day of the survey, information on each patient 80 years or older hospitalized in the service will be collected:

* Patient Data: date of birth, sex, status. The patient identification data (name, surname, address) will not be collected.
* Patient History: date of last hospitalization, life, cardiovascular risk factors, cardiovascular and non cardiovascular history, date of last hospitalization, life
* Circumstances of admission: course of care before admission, admission to intensive care unit or hospital unit classical primary diagnosis and diagnosis (s) partner (s)
* Initial assessment: treatment admission, major hemodynamic, electrocardiographic and biological
* Regarding the current hospitalization: diagnosis already implemented or planned (echocardiography, angiography, electrophysiological study, etc ...), therapeutic methods already implemented or planned angioplasty, percutaneous valve intervention, conventional or biventricular stimulation, cardiac surgery, medication
* Become of the patient after hospitalization
* The clinician's subjective impressions about the condition of the patient and monitoring recommendations
* Assessment of addiction: ADL Scale

No monitoring of patients is contemplated.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 80 years or more
* Patient present in a cardiology service in the morning (8:00 to 12:00) the day of the survey
* Admission to the service took place on the survey day or in the 15 days preceding the survey.

Exclusion Criteria:

* Patient with age <80 years.
* Patient who have expressed a refusal to participate in the study

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 80 years and older and hospitalized in a cardiology department which participate in this study.
Sampling Method: Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients for which national guidelines were followed | 1 day
  Evaluate clinical practice and particularly the monitoring of recommendations of international scientific societies in the population of very elderly (≥ 80 years)

SECONDARY OUTCOMES:
Percentage of patients aged 80 and older hospitalized in the university and non university | 1 day
  Better understand the demographics of cardiology services in France (Demography)

CONTACTS AND LOCATIONS:
Locations (1):
- Lariboisiere Hospital, Paris, France

REFERENCES:
- [Result] Moubarak G, Ernande L, Godin M, Cazeau S, Vicaut E, Hanon O, Zuily S, Tournoux F, Danchin N, Derumeaux G, Mechulan A. Impact of comorbidity on medication use in elderly patients with cardiovascular diseases: the OCTOCARDIO study. Eur J Prev Cardiol. 2013 Aug;20(4):524-30. doi: 10.1177/2047487312444235. Epub 2012 Mar 23. PMID 22447578